The Ohio State University Combined Consent to Participate in Research and HIPAA Research Authorization

2

1

SPASM: Randomized, Sham Controlled Trial of Dorsal Root

Study Title: Rhizotomy Stereotactic Radiosurgery versus Standard of Care for Specific Associated with Stroke Spinel Cord Injury & Carebral

Spasticity Associated with Stroke, Spinal Cord Injury & Cerebral

**Palsy** 

Principal Investigator: Evan M. Thomas, MD, PhD

**Sponsor:** Varian Medical Systems

4 5

6

7 8 • This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.

9 10 11

12

13

• Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.

14 15 16

You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.

17 18

19

20

21

• You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

222324

25

#### **Key Information About This Study**

The following is a short summary to help you decide whether or not to be a part of this study. More detailed information is listed later in this form.

262728

29

30

31

32

This study is being done to determine the safety and effectiveness of high dose focused radiation to a part of your spine called the spinal dorsal root using a technique called stereotactic radiosurgery (SRS) in patients with spasticity. If you agree to participate in the study, you will be randomly assigned to either receive radiosurgery or not to receive radiosurgery. As part of your participation in the study, you will be asked to complete follow-

up visits at 2, 6, 12, and 24 months. If you are randomized to the group without radiosurgery,

you will be allowed to crossover to the group receiving radiosurgery after your 6 month visit if you desire.

#### 1. Why is this study being done?

This study will evaluate the safety and effectiveness of high-dose focused radiation to the spinal dorsal root using a technique called stereotactic radiosurgery (SRS) in patients with spasticity. Stereotactic radiosurgery is the precise high dose application of radiation to a small area. A dorsal root rhizotomy is the intentional damage or change to the root of the nerve coming out of the spinal cord that carries sensory information. In patients with spasticity, this is the part of the nerve that sends too much signal to the spinal cord and causes heightened reflexive spasticity. Radio surgical rhizotomy is noninvasive and uses focused radiation to attempt to change the function of the nerve without destroying it. The purpose of this study is to see if using 1 treatment session of SRS for spasticity is safe and helps your spasticity.

You are being asked to take part in this study because you have spasticity that is still present despite medical or other interventional management.

#### 2. How many people will take part in this study?

It is anticipated that up to 25 patients will take part in this study at Ohio State.

# 3. What will happen if I take part in this study?

#### Before you begin the study:

The following will take place to find out if you can be in the study. These exams, tests, or procedures are sometimes part of regular medical care. If you have recently had them done, they may not need to be repeated. Your medical record will be reviewed by the study doctor to determine which tests and procedures will be needed.

• A physical examination

 • Your medical history will be collected, and you will complete an interview that includes questions about your past and current health.

• Evaluation of your spasticity and its effects on your quality of life. You will be assessed and asked questions. Your spasticity and its effect on your quality of life will be assessed.

• Evaluation of your ability to carry out daily activities. You will be asked questions about what type of daily activities you can do.

• Imaging of your spine with Magnetic Resonance Imaging (MRI) and Computer Tomography (CT) imaging.

IRB Protocol Number: 2022H0425 IRB Approval date: 9/22/2023 Version: 1.0

- o MRI scans create images of the body using a strong magnet and radio waves. You will be asked to remove all metal objects from your person before entering the scanning room and may be asked to remove clothing and put on a hospital gown or scrubs. During the MRI scan, you will lie on a table and be confined toa small space inside a cylindrical machine (tube). The MRI will take about 1 hour. Although you will be asked not to move or talk during the MRI procedure, you will be able to communicate with the MRI Technologist by pressing a call button that will be within your reach. The Technologist will observe you during the entire time that you are in the MRI scanner.
- o CT is a way to make x-ray images of the inside of the body. The CT scanner is a doughnut-shaped machine that uses x-rays to create pictures that show structures inside your body more clearly than regular x-ray pictures. During the procedure, a technologist will take you into the CT scan room where you will lie down on the inside of the CT machine. During the study, you will be asked to hold your breath so that the pictures will not be blurred. The machine will make some noise, and the table will move during the scan. The scan will take about 1 hour.
- Electromyogram (EMG) and nerve conduction velocity (NCV) testing to see how your muscles and nerves are working. This will only be done if it is part of your standard of care treatment. If you are not undergoing EMG and NCV as part of your regular medical treatment, it will not be done separately for this study.
  - EMG is a procedure that assesses the health of your muscle and nerve cells by measuring the electrical activity of your muscles as they move. An EMG measures these impulses through a needle, which acts as an electrode, injected into the muscle tissue. The EMG will take approximately 30-90 minutes.
  - A NCV test measures how fast electrical impulses move through your nerves. During the test, your nerve will be stimulated, and the nerve activity recorded with electrode patches attached to your skin. The NCV will take approximately 30-90 minutes.

#### **During study treatment:**

- You will undergo another CT scan. This CT scan is used to design a radiosurgery treatment plan. It will take approximately 1 hour.
- You will be randomly assigned (like flipping a coin) to either the treatment group or the "sham" group. There is a 50/50 chance of being in either group. You will not be able to choose what group you are assigned to, and you will not know what group you are assigned to.
  - Regardless of which group you are assigned to; you will be asked to lie on the treatment table and a device will rotate around you. This will take approximately 30-90 minutes.

IRB Protocol Number: 2022H0425
IRB Approval date: 9/22/2023
Version: 1.0

o **If you are assigned to the treatment group,** you will receive a radiosurgery treatment to one or more of your affected nerve roots. The device rotating around you will emit invisible, high-energy x-rays.

o **If you are assigned to the "sham" group,** you will not receive treatment. The device rotating around you will not emit x-rays.

124125

120

121122

123

#### After you are finished with treatment:

126 127 128

129

130

131

132

133

134

135

136

137

You will be asked to complete follow-up visits at 2 months, 6 months, 12 months, and 24 months after treatment. Each follow-up visit will take 45 - 90 minutes and include the following:

- Physical examination
- Evaluation of your spasticity and its effects on your quality of life
- Evaluation of your ability to carry out daily activities
- Imaging of your spine with MRI and CT imaging
- EMG and NCV testing (only at the 6 month visit). This will only be done if it is part of your standard of care treatment. If you are not undergoing EMG and NCV as part of your regular medical treatment, it will not be done separately for this study.

138139140

141

142

In addition, the researchers will access your medical records to obtain information related to your demographics, medical history, and spasticity. If you have had photos taken as part of your standard of care spasticity assessment, these may be obtained from your medical records as well.

143144145

If you are randomized to the group without radiosurgery, you will be allowed to crossover to the group receiving radiosurgery after your 6 month visit if you desire.

146147148

#### 4. How long will I be in the study?

149150

You will be in the study for 24 months after treatment.

151152

# 5. Can I stop being in the study?

153154

155

156

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

157158

# 6. What risks, side effects or discomforts can I expect from being in the study?

159160161

163

#### **Risks related to the SRS Treatment:**

162 <u>Likely:</u>

• Dullness or changing of sensation in the area being treated for spasticity

Page 4 of 12

Changes in muscle spasm patterns in the area being treated for spasticity

164165166

167

168

169

170

#### **Less Likely:**

- Reddening of the skin in the area treated with radiation
- Pain at the site of radiation treatment
- Swelling around the area of the treatment
- Scar tissue formation in the area of treatment
- Changes in how your limb being treated feels

171172173

#### Rare but potentially serious:

- Injury to the spinal cord near the area receiving treatment
- Necrosis or injury to skin or soft tissue near the treatment area

175176177

178

179

180

181

182

183

184

185

186

187

174

#### **Information for Women of Childbearing Potential**

If you are pregnant, you cannot take part in this study. You should not become pregnant if you decide to take part because the radiation can affect an unborn baby. This study may be harmful to a nursing infant or an unborn child. If you are unwilling to use adequate birth control measures to prevent pregnancy, you cannot participate in this study. Reliable methods of birth control are considered to be: abstinence (not having sex), intrauterine device (IUD), tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts). An acceptable, although less reliable method involves the careful use of condoms and a spermicidal foam or gel and/or a cervical cap or sponge. It is important you understand that you need to use birth control while on this study and for 6 months after treatment ends. If you suspect that you are pregnant or if you become pregnant while you are on this study, you must tell your doctor immediately.

188 189 190

191

192

193

194

195

#### **Radiation Risks**

This research study involves exposure to radiation from CT scans of your spine and from the radiosurgical procedure. This radiation exposure is for research purposes only. The total amount of radiation that you will receive in this study is about 535.4 mSv and is approximately equivalent to a whole body exposure of 89 years of exposure to natural background radiation. Most of this radiation is concentrated within the nerve root being treated. The exposure to the body as a whole is much less.

196 197 198

199

200

201

#### **Loss of Confidentiality**

There is a risk of loss of confidentiality, but many precautions will be taken to protect your information.

202203

# 7. What benefits can I expect from being in the study?

204205206

207

You may or may not benefit from taking part in this study. SRS for spasticity may be effective in treating spasticity. However, there is no proof of this yet.

IRB Protocol Number: 2022H0425
IRB Approval date: 9/22/2023

Version: 1.0

208209

The information gained from this study will help doctors learn more about SRS as a treatment for spasticity, which could help other patients in the future.

210211212

#### 8. What other choices do I have if I do not take part in the study?

213214

Your other choices include getting the current standard of care treatment for spasticity without being in a study or taking part in another, unrelated study that may be available.

215216217

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

218219220

#### 9. What are the costs of taking part in this study?

221222

The costs of your standard medical care will be billed to you and/or to your insurance company in the usual manner.

223224225

You and your health insurance plan are responsible for all routine costs associated with this study. Routine costs are costs that are covered by Medicare in connection with studies such as this one, even if Medicare is not your insurance provider.

227228229

230

231

232

233

226

All routine costs will be billed to your health insurance plan, but there is no guarantee that your health insurance plan will cover all routine costs. Even where such insurance coverage is provided, you may still have to pay some costs such as copayments, coinsurance, or deductibles for the covered items or services. You should contact your health plan to discuss its coverage policy for items or services provided during a research study.

234235236

#### 10. Will I be paid for taking part in this study?

237238

You will not receive payment for participating in this study.

239240

# 11. What happens if I am injured because I took part in this study?

241242243

244

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

245246

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

248249

247

# 12. What are my rights if I take part in this study?

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

254255256

257

252

253

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

258259260

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

261262263

264

265

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

266267268

269270

## 13. Will my de-identified information be used or shared for future research?

Yes, it may be used or shared with other researchers without your additional informed consent.

271272273

#### 14. Will my study-related information be kept confidential?

274275

276

277

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

278279280

Also, your records may be reviewed by the following groups (as applicable to the research):

281282

• Office for Human Research Protections or other federal, state, or international regulatory agencies;

283 284

• U.S. Food and Drug Administration;

285286

• The Ohio State University Institutional Review Board or Office of Responsible Research Practices;

287288

The sponsor supporting the study, their agents or study monitors; and
Your insurance company (if charges are billed to insurance).

289 290

If we find information that significantly impacts your health, we will share it with you. This includes information as to the efficacy of the treatment or potential adverse effects of treatment.

292293294

295

291

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At

IRB Protocol Number: 2022H0425
IRB Approval date: 9/22/2023

Version: 1.0

| 296 | most, the website will include a summary of the results. | You can search the website at |
|---|---|---|
| 297 | any time. | |

298299

# 15. HIPAA AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

300301

#### I. What information may be used and given to others?

302303

• Past and present medical records;

304

• Research records;

305 306

• Records about phone calls made as part of this research;

307

Records about your study visits;
Information that includes personal identifiers, such as your name, or a number

308 309

associated with you as an individual;Information gathered for this research about:

310 311

Physical exams

Laboratory, x-ray, and other test results

Diaries and questionnaires

313 314

• Records about the study device

315316

#### II. Who may use and give out information about you?

317318

Researchers and study staff.

319320

# III. Who might get this information?

321 322

- The sponsor of this research. "Sponsor" means any persons or companies that are:
- working for or with the sponsor; or

323324

• owned by the sponsor.

325326

Authorized Ohio State University staff not involved in the study may be aware that you are participating in a research study and have access to your information;
If this study is related to your medical care, your study-related information may be

placed in your permanent hospital, clinic, or physician's office record;

327328329

IV. Your information may be given to:

330331332

333

335

- The U.S. Food and Drug Administration (FDA), Department of Health and Human Services (DHHS) agencies, and other federal and state entities;
- Governmental agencies in other countries;
  - Governmental agencies to whom certain diseases (reportable diseases) must be reported; and

The Ohio State University units involved in managing and approving the research study including the Office of Research and the Office of Responsible Research Practices.

339 340

337

338

#### V. Why will this information be used and/or given to others?

341

342 • To do the research:

343

344

• To study the results; and

345

• To make sure that the research was done right.

346 347

# VI. When will my permission end?

348 349

There is no date at which your permission ends. Your information will be used indefinitely. This is because the information used and created during the study may be analyzed for many years, and it is not possible to know when this will be complete.

351 352 353

350

# VII. May I withdraw or revoke (cancel) my permission?

354 355

356

357 358

359

360

Yes. Your authorization will be good for the time period indicated above unless you change your mind and revoke it in writing. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the researchers. If you withdraw your permission, you will not be able to stay in this study. When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

361 362 363

#### VIII. What if I decide not to give permission to use and give out my health information?

364 365 366

367

368

Then you will not be able to be in this research study and receive research-related treatment. However, if you are being treated as a patient here, you will still be able to receive care.

369 370

# IX. Is my health information protected after it has been given to others?

371 372

There is a risk that your information will be given to others without your permission. Any information that is shared may no longer be protected by federal privacy rules.

373 374 375

# X. May I review or copy my information?

376 377

Signing this authorization also means that you may not be able to see or copy your studyrelated information until the study is completed.

IRB Protocol Number: 2022H0425 IRB Approval date: 9/22/2023

Version: 1.0

380 381

## 16. Who can answer my questions about the study?

382 383

For study questions, concerns, or complaints, to withdraw consent and HIPAA authorization, or if you feel you have been harmed as a result of study participation, you may contact **Evan Thomas, MD at 614-293-8415.** 

385386387

388

384

For questions related to your privacy rights under HIPAA or related to this research authorization, please contact the HIPPA Privacy officer located at 650 Ackerman Rd Columbus, OH 43210, 614-293-4477 or 614-293-7672.

389390391

392

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

393394395

If you are injured as a result of participating in this study or for questions about a study-related injury, you may contact **Evan Thomas, MD at 614-293-8415.** 

396397398

399

400

401

402

Dr. Evan Thomas, a researcher helping to perform this study, is a paid consultant for Varian Medical Systems, Inc., the manufacturer of the devices being tested. A conflict of interest committee at Ohio State has reviewed this information and determined that Dr. Thomas's involvement presents no additional significant risk to the study's participants. Any questions about this information can be answered by Dr. Joshua Palmer, (614) 293-8415

| Signing the consent form | |
|---|---|
| | s form and I am aware that I am being asked to<br>he opportunity to ask questions and have had the<br>gree to participate in this study. |
| I am not giving up any legal rights by signing combined consent and HIPAA research authorized to the combined consent authorized to the combined con | |
| Printed name of participant | Signature of participant |
| | Date and time AN |
| Printed name of person authorized to consent for | Signature of person authorized to consent for participan (when applicable) |
| participant (when applicable) | |
| participant (when applicable) Relationship to the participant | Date and time |
| Participant (when applicable) Relationship to the participant Optional photo consent: Please check one the research team to collect any available phrecord for the research. | Date and time of the boxes below to indicate whether you allowed a related to your spasticity from your medicate. |
| Participant (when applicable) Relationship to the participant Optional photo consent: Please check one the research team to collect any available phrecord for the research. I agree to have photos collected from my | Date and time of the boxes below to indicate whether you allow notos related to your spasticity from your medicate. |
| Participant (when applicable) Relationship to the participant Optional photo consent: Please check one the research team to collect any available phrecord for the research. I agree to have photos collected from my | Date and time of the boxes below to indicate whether you allowed a second to your spasticity from your medicate whether you allowed a second to your spasticity from your medicate whether you allowed a second to your spasticity from your medicate whether you allowed a second to your spasticity from your medicate whether you allowed to your spasticity from your medicate your medicate whether you allowed to your spasticity from your medicate your medic |
| Relationship to the participant Optional photo consent: Please check one the research team to collect any available phrecord for the research. I agree to have photos collected from my I DO NOT agree to have photos collected Investigator/Research Staff I have explained the research to the participation. | Date and time of the boxes below to indicate whether you allowed notos related to your spasticity from your medical medical records for this research. ed from my medical records for this research. |
| Relationship to the participant Optional photo consent: Please check one the research team to collect any available phrecord for the research. I agree to have photos collected from my I DO NOT agree to have photos collected Investigator/Research Staff I have explained the research to the participation signature(s) above. There are no blanks in the state of the participation of th | Date and time of the boxes below to indicate whether you allowed a second to your spasticity from your medicate whether you allowed a second to your spasticity from your medicate whether you allowed a second to your spasticity from your medicate whether you allowed a second to your spasticity from your medicate whether you allowed to your spasticity from your medicate your medicate whether you allowed to your spasticity from your medicate your medic |

IRB Protocol Number: 2022H0425 IRB Approval date: 9/22/2023 Version: 1.0

| Printed name of witness | Signature of witness | Signature of witness |
|-------------------------|----------------------|----------------------|
| | Date and time | AM/PM |
| Printed name of witness | Signature of witness | |
| | Date and time | AM/PM |